CLINICAL TRIAL: NCT02842879
Title: Outpatient Versus Inpatient Cervix Priming With Foley Catheter
Brief Title: Outpatient Foley Cervix Priming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Catarina Policiano, Dr. Catarina Policiano, Hospital de Santa Maria, Portugal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SantaMariaPortugal
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Outpatient Mechanical Cervix Priming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Foley cervix priming (Experimental): Patients randomized to outpatient cervix priming will have the insertion of the catheter in the same conditions defined by the Department protocol for inpatient cervix priming. They will be discharged after a reassuring cardiotocogram following the introduction of the Foley catheter. When discharged, the patients will be instructed to apply manual traction to the catheter every 6 hours and they will be given a written document with all the information that should bring them back to hospital.
  Interventions: Other: Outpatient Foley cervix priming
- Inpatient Foley cervix priming (No Intervention): The introduction of a deflated catheter (Foley catheter nº 16F) through the outer cervix orifice is preceded by iodine disinfection of the cervix. The intracervical catheter is distended with 40mL of a saline solution. The end of the catheter is taped to the medial portion of the thigh and manual traction is applied to the catheter every 6 hours. If it is not spontaneously extruded it is removed after 24h. Cervix priming occurs in an inpatient setting.

INTERVENTIONS:
Other: Outpatient Foley cervix priming — Outpatient setting for cervix priming with Foley catheter
  Arms: Outpatient Foley cervix priming

SUMMARY:
The aim was to conduct a non-blinded prospective randomized study at a tertiary hospital. Inclusion criteria: term pregnancy with a single fetus in cephalic presentation, Bishop score < 6, gestational age > 41 weeks or medical indication for induction of labor.

Patients will be randomized to outpatient or inpatient cervix priming with Foley catheter.

The primary outcome will be to compare the variation of Bishop score (difference between Bishop score before and after application of Foley catheter) between outpatient and inpatient groups. Secondary comparisons include: mode of delivery, Foley catheter application-to-delivery time, inpatient time, sequential use of prostaglandins, infection and maternal pain.

ELIGIBILITY:
Inclusion Criteria:

* women with a single fetus in cephalic presentation
* Bishop score < 6
* Gestational age > 41 weeks or medical indication for induction of labor submitted to cervix priming with Foley catheter

Exclusion Criteria:

* women with a fetus in noncephalic presentation
* an indication for elective cesarean delivery
* spontaneous labor
* hydramnios (amniotic fluid index ≥ 25)
* nonreassuring cardiotocogram
* multiple pregnancy
* rupture of membranes
* active vaginal bleeding
* indication for prophylaxis of Streptococcus group B infection
* HIV infection
* cervical injury
* previous cesarean section with recurrent indication

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
variation of bishop score (difference between bishop score before and after application of foley catheter) | up to 24 months

SECONDARY OUTCOMES:
mode of delivery | up to 24 months
induction-to-delivery time | up to 24 months
maternal pain evaluated by visual analog scale for pain | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Policiano, MD, Principal Investigator — Hospital de Santa Maria, Centro Hospitalar Lisboa Norte

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803
- [Derived] Policiano C, Pimenta M, Martins D, Clode N. Outpatient versus inpatient cervix priming with Foley catheter: A randomized trial. Eur J Obstet Gynecol Reprod Biol. 2017 Mar;210:1-6. doi: 10.1016/j.ejogrb.2016.11.026. Epub 2016 Nov 27. PMID 27923165